CLINICAL TRIAL: NCT07142512
Title: A Dyadic Coping Strategy to Enhance Step Prescription Effects in Type 2 Diabetes: a Bayesian Adaptive Basket Randomized Controlled Trial
Brief Title: Helping Couples Communicate Better: Does This Help Persons With Type 2 Diabetes Respond Better to a Step Count Prescription?
Acronym: PartnerStepT2D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Diabetes Canada (Other)
Responsible Party: Principal Investigator, Kaberi Dasgupta, MD, MSc, FRCP (C), Senior Scientist, Professor of Medicine, Physician, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OG-323-5723-KD
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Partner; Spouse; Wife; Husband; Step counts; Step targets; Hemoglobin A1C; Couple counseling; Dyadic coping
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: As discussed in the detailed description of the trial, this is a a Bayesian adaptive basket randomized controlled trial. There are 4 prespecified subgroups (high marital quality- lower marital quality, both partners with obesity- one or neither with obesity).
Masking Description: The technicians who perform the assays (hemoglobin A1C, lipid profiles) are masked to study arm. Steps/day measurements are captured through step counting devices. Blood pressure and weight are assessed through automated devices.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step Count tracking and goals alone (Active Comparator): We will provide this active comparator arm with weekly step count goals and a step counter for the 24 week study period. We provide further details in the description of the intervention with the same title.
  Interventions: Behavioral: Step Count tracking and goals
- Step Count tracking and goals with dyadic coping intervention (Experimental): This arm will receive the same step tracking and goal intervention described for the active comparator but will additionally participate in the dyadic coping intervention.
  Interventions: Behavioral: Step Count tracking and goals; Behavioral: Dyadic coping intervention

INTERVENTIONS:
Behavioral: Step Count tracking and goals — We will provide participants and partners with Fitbits for the duration of the trial. After one week of step counting, the next week target will be to increase by 500 steps/day if baseline < 5000 steps/day; increase by 750 steps/day if baseline 5000 to 7,500 steps/day; and increase by 1,000 steps/day if baseline > 7,500 steps/day). Each week thereafter, study staff will pull the step data and apply an algorithm to generate new targets for the next week. In our algorithm, subsequent targets are higher if the participant exceeds prior week targets, and lower/unchanged if below target. This is similar to the algorithm we used in our trial ACTIVE PATIENT GDM (Dasgupta K, Chan D, Bond R, Garfield N, Coolen J, Halperin IJ, Peters TM, et al. Step and weight tracking with targets and coaching interventions in gestational diabetes: A randomized factorial feasibility trial. Diabetes Res Clin Pract. 2025 Jun;224:112241. doi: 10.1016/j.diabres.2025.112241. Epub 2025 May 9. PMID: 40349846.)
Behavioral: Dyadic coping intervention — Couples will participate in 8 one-hour coaching sessions over 12 weeks (virtual, in-person, or a combination, as preferred). The sessions aim to enhance the couple's understanding of how they influence each other. Both couple members will explore their preferences in terms of ways of communicating and supporting one another's goals. We will use changes in steps as a context to explore how partners can effectively support and "coach" each other without without eliciting behavioural reactance. We will use are goal setting, action planning, self-monitoring, graded tasks, social environment restructuring, and social support. The coaches will be psychology students. They will receive structured training on the coaching strategy from a licensed mental health professional. We will record the sessions for fidelity and quality assurance purposes. All coaches will meet weekly with the supervising licensed mental health professional.
  Arms: Step Count tracking and goals with dyadic coping intervention

SUMMARY:
Being active is one way to reach better blood sugar control and heart health in type 2 diabetes. The investigators developed a strategy to help people with type 2 diabetes walk more. They track their steps with a step counter and set targets with their doctor through a kind of 'step prescription.' While this strategy helps people increase their physical activity, it can be useful to have support besides the clinic visits. Their partner might be a good person to help.

Partners often have similar activity levels. Partners of people with type 2 diabetes are also more likely to develop type 2 diabetes. There are good reasons to work together! However, not all partners communicate in a way that helps them work together effectively. The investigators are going to give a step counter and step prescriptions to a large group of people with type 2 diabetes. The partners will also receive counters and step prescriptions. Half of the couples will be randomized (assigned to a group based on something equivalent to a coin toss) to participate in online or in-person sessions with a counselor. They will work together to figure out how to communicate more kindly and effectively. The investigators will see if the people with these sessions wind up having higher steps and better sugar control than the people who do not. To figure out in which types of couples the strategy works, The investigators will also divide the couples into groups based on the type of marriage that they have (figured out through a questionnaire) and body size. The investigators will see if the counseling strategy helps in both 'high' and 'low' quality relationships and if couples where both partners have extra weight respond differently to the strategy than other couples. During the trial, if The investigators see that the strategy is not working well in one particular group of people, The investigators may recruit fewer in this group and more in the others. The investigators will do this in consultation with specialized statisticians who will look at the data at specific points in time. This is a way of making sure that the investigators are testing the right strategy in the right group, increasing the 'efficiency' and relevance of the study.

DETAILED DESCRIPTION:
Persons with type 2 diabetes (T2D; henceforth, persons with diabetes, PWD) face personal (e.g., time pressure, competing priorities), social (e.g., food commercialization, employment and leisure digitization, inequity), and psychological (e.g., distress) challenges in addressing key behaviours that affect glycemic control, cardiometabolic profiles, and T2D complications. These behaviours include excess calorie intake, consumption of low nutrient quality food and beverages, low physical activity, high sedentary time, and poor sleep habits. Partners are potential assets in supporting positive health behaviour change. They often share lifestyle behaviours and may be at risk for similar outcomes. However, some couples may need adjustments in communication and relational dynamics, to work collaboratively towards healthier behaviours.

The investigators will examine a dyadic coping intervention that the investigators have developed, in terms of its efficacy in stimulating positive behaviour changes in PWD who have partners. In this study, the behaviours that the investigators will specifically focus on are low physical activity and high sedentary time. The investigators will apply an adapted version of our trial-tested SMARTER step count prescription strategy, now integrated into Diabetes Canada guidelines. The investigators will compare its effects alone vs. combined with our dyadic coping intervention, on step counts in persons with type 2 diabetes and their partners. The investigators will also examine changes in hemoglobin A1C in the index participant with type 2 diabetes. In the spirit of precision medicine and statistical efficiency, the investigators will apply an adaptive basket trial design to delineate in which profiles (marital quality [Couples Satisfaction Index-16 divided as score < 61 vs. 61 or higher] , concordance for BMI > 30 kg/m2 vs. not) the dyadic coping intervention is likely to demonstrate efficacy. Couples with higher marital quality and/or shared impact of less healthy behaviours or environments (as reflected by concordance in excess weight) may experience stronger impact of the intervention.

In addition to the outcomes described below, the investigators will assess participant perspectives regarding the dyadic coping intervention. Through a descriptive qualitative approach (exit in-depth interviews), the investigators will explore experiences of couples in the dyadic coping intervention arm. The investigators will use a semi-structured interview approach, using the guide that the investigators have developed. The investigators will interview both members of the couple together, by telephone. The investigators will continue sampling until saturation of themes occurs. The investigators will audio record and transcribe the interviews. Two trained investigators will read and code for themes. Data coding/organisation will be facilitated by Dedoose Version 7.0.23 and NVivo analysis software. Data analysis will be informed by thematic analyses.

What did the participant like about the approach? (coaching, step monitoring, goals) What did the participant not like? How would the participant improve the approach? How were the number of coaching sessions? Too many? Too few? How was the length of the coaching sessions? Too long? Too short?

ELIGIBILITY:
Inclusion Criteria:

* (i) Index participant has T2D;
* (ii) Index participant 45 years of age or older;
* (iii) Index participant and partner: Co-habiting with a partner (same or different sex) for two or more years;
* (iv) Index participant and partner: Absence of gait difficulties or other co-morbid conditions that impede walking in the index participant;
* (v) Willingness to complete an audiovisual recording of a conversation between the couple members to capture couple communication styles
* (vi) Index participant and partner Smartphone and Internet access.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in steps/day | The primary outcome is at 24 weeks and a secondary outcome will be at 12 weeks (midpoint)
  Difference between mean baseline (week 1) and final (week 24) steps/day; daily steps are automatically uploaded to a secure cloud-based server and pulled by our research team for weekly goals and outcome assessment. We require at least 4 days of measurement. If sufficient days are not captured in week 1, we may compute based on the earliest of weeks 2 through 4 that includes sufficient data. If sufficient days are not captured in week 24, we may compute based on the latest of weeks 20 through 24 that includes sufficient data.

SECONDARY OUTCOMES:
Change in A1C | 24 weeks
  We will assess the difference between hemoglobin A1C (measure of glycemic control) between baseline and final assessment.
Change in insulin resistance | 24 weeks
  We will assessed fasting insulin and fasting glucose levels at baseline and following the intervention. We will use these values to compute the Homeostatic Model Assessment-Insulin Resistance [HOMA-IR] measure.
Change in systolic blood pressure | 24 weeks
  We will evaluate the change in systolic blood pressure between baseline and final assessments. This will be based on the average of 5 sequential automated oscillometric blood pressure monitor-assessed values.
Total steps | 24 weeks
  We will sum total steps over the study period.
Dyadic coping | 24 weeks
  We assess this through the common dyadic coping subscale (5 questions) of the Dyadic coping inventory (each question with 5 Likert scale options). We will look at the difference in total score between baseline and final assessments.
  Reference: Bodenmann G, Arista LJ, Walsh KJ, et al. Dyadic Coping Inventory. In: Lebow J, Chambers A, Breunlin DC, editors. Encyclopedia of Couple and Family Therapy. Cham: Springer International Publishing; 2018. p. 1-5.

OTHER OUTCOMES:
Change in body mass index (BMI) | 24 weeks
  We will assess the difference in BMI between baseline and final assessments. We will use measured weight (digital scale) and height (stadiometer) values to compute BMI as weight in kilograms divided by height in meters squared.
Change in marital quality | 24 weeks
  In both index participants and their partners, we will assess the difference between questionnaire-assessed marital quality during the first week and the final week of the intervention. We will use the Couples Satisfaction Index (16 item version; score range 0 to 80).
  Reference: Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007;21(4):572-83.
Change in high-density lipoprotein cholesterol (HDL) | 24 weeks
  We will evaluate the difference in HDL between baseline and final assessments.
Change in self-efficacy for physical activity | 24 weeks
  We are using reactions to the following questions to assess physical activity-related self-efficacy (5-point Likert scale- strong disagree, disagree, neutral, agree, strongly agree): I possess the skills to do regular physical activity over the next 6 months if I wanted to. I have the ability to do regular physical activity over the next 6 months if I wanted to. I am confident that I am capable of engaging in regular physical activity if I had to.
  We will use similar questions to assess perceptions of the partner's self-efficacy, substituting 'my partner' for 'I' in the above series of questions. Both the index participant and the partner participant will answer both series of questions.
  Reference: Burrell AMG, Allan JL, Williams DM, et al. What do self-efficacy items measure? Examining the discriminant content validity of self-efficacy items. British journal of health psychology. 2018;23(3):597-611.
Low density lipoprotein cholesterol (LDL) | 24 weeks
  We will assess the difference between LDL values at baseline and final assessments. LDL is calculated from total cholesterol, HDL, and triglyceride values.
Change in percent body fat | 24 weeks
  We will assess the difference in percent body fat between baseline and final assessments. We will use the Tanita BF-350 Body Composition Analyzer for Bioelectrical Impedance Analysis (BIA).
Change in diastolic blood pressure | 24 weeks
  We will evaluate the change in diastolic blood pressure between baseline and final assessments. This will be based on the average of 5 sequential automated oscillometric blood pressure monitor-assessed values.
Change in exercise-related motivation | 24 weeks
  We will examine change in intrinsic and integrated motivation using changes in the intrinsic and integrated regulation subscales of the Behavioural Regulations in Exercise Questionnaire (18 questions each with a 0 to 4-point Likert scale).
  Reference: Markland D, Tobin V. A modification to the Behavioural Regulation in Exercise Questionnaire to include an assessment of amotivation. Journal of Sport & Exercise Psychology. 2004;26(2):191-6.
Change in diabetes distress | 24 weeks
  We will assess the difference in diabetes distress between baseline and final assessments using the Diabetes Distress Scale. The index participant will complete the version for people living with type 2 diabetes (17 potential problem areas; scored on Likert scale 1 through 6 for related distress). Partners who have type 2 diabetes will also complete this version. All partners will complete the partner version of the Diabetes Distress Scale (2 potential problem areas; Likert scale 1 through 6).
  Reference: Polonsky W, Fisher L, Earles J, et al. Assessing psychosocial distress in diabetes: Development of the diabetes distress scale. Diabetes Care. 2005;28(3):626-31.
Change in degree of depressed mood | 24 weeks
  We will assess the change in depressed mood between baseline and final assessment as captured by the change in score on the Center for Epidemiologic Studies Depression Scale (CES-D).
  Reference: Radloff LS. The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977;1(3):385-401.
Change in dietary habits | 24 weeks
  We will assess the difference in healthy eating between baseline and final assessments using the total score of the Starting the Conversation on Diet questionnaire (8 items; each with 3 categories related to frequency [first 7] or amount [last item] of intake- fast food, fruit, vegetables, sweetened beverages, beans/chicken/fish, chips/crackers, desserts/sweets, margarine/butter/fat).
  Reference: Paxton AE, Strycker LA, Toobert DJ, et al. Starting the conversation performance of a brief dietary assessment and intervention tool for health professionals. Am J Prev Med. 2011;40(1):67-71.

CONTACTS AND LOCATIONS:
Overall Officials: Kaberi Dasgupta, MDCM, MSc, FRCPC, Principal Investigator — Research Institute of the McGill University Health Centre; Jean-Philippe Gouin, PhD, Principal Investigator — Concordia University, Montreal; Shirin Golchi, PhD, Principal Investigator — McGill University
Locations (3):
- Canada (3):
  - St. Mary's Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
Following completion of all trial procedures, we will perform the analyses and write the manuscript reporting the trial results. We may then consider data sharing on a case by case basis, subject to review of analysis plans, ethics review, and formal agreements.